CLINICAL TRIAL: NCT06791265
Title: Computer-guided Versus Conventional Eminectomy for Treatment of Recurrent Temporomandibular Joint Dislocation
Brief Title: Computer-guided Versus Conventional Eminectomy
Acronym: Computer-guide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Amr Gibaly, Associate Professor of Oral and Maxillofacial Surgery, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16
Record Dates: First submitted 2025-01-10; First posted 2025-01-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: TMJ - Dislocation of Temporomandibular Joint

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Eminectomy (Active Comparator): computer-guided osteotomy
  Interventions: Device: Guided Eminectomy
- Free hand Eminectomy (Active Comparator): conventional osteotomy
  Interventions: Procedure: Free hand Eminectomy

INTERVENTIONS:
Device: Guided Eminectomy — The patients will be subjected to computer-guided osteotomy utilizing a virtually preplanned cutting guide
  Arms: Guided Eminectomy
Procedure: Free hand Eminectomy — The patients will be subjected to a free-hand Eminectomy utilizing the routine surgical technique
  Arms: Free hand Eminectomy

SUMMARY:
Dislocation of temporomandibular joint (TMJ) is a pathologic condition in which the patient suffers non-self limiting hypermobility in the joint due to the displacement of mandibular condyle outside its position within the glenoid fossa. Although lateral and posterior dislocation is mentioned in literature, Anteromedial position is the most common. In this condition, the condyle is stuck beyond the articular eminence anteriorly in a non-functional position.

DETAILED DESCRIPTION:
TMJ dislocation occurs in different forms, acute dislocation as a result of trauma or excessive opening, chronic dislocation as a result of capsule laxity due to prolonged disarticulation, and finally recurrent dislocation. Recurrent dislocation is a repeated sporadic acute TMJ dislocation. Unlike chronic dislocation, the mandibular condyle is located in its normal position between dislocation episodes. Recurrent TMJ dislocation treatment modalities can be organized according to the stability factor into ligaments alteration, musculature alteration, and bony anatomy alteration. Nonsurgical/minimally invasive and surgical/invasive therapies have been used. Conservative modalities are usually used before invasive modalities, yet surgical modalities are still superior to non surgical modalities due to its higher success rate. Eminectomy is one of the widely used surgical procedures to manage recurrent dislocation. It is considered as a "rescue procedure" by many surgeons

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an age range of 18-60 years, males and females, with bilateral dislocation o
2. Medically free

Exclusion Criteria:

medically compromised patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Dislocation recurrence | 6 months
  The recurrence will be investigated for ocuurence in the followups

SECONDARY OUTCOMES:
Maximum interincisal opening (MIO) | 6 months
  maximum mouth opening will be measured in followups
Accuracy of the digital workflow | One week postoperative
  The accuracy of the work flow will be assessed by superimposing the CBCT scans

CONTACTS AND LOCATIONS:
Locations (1):
- Amr Gibaly, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No